CLINICAL TRIAL: NCT01767961
Title: A Pilot Study Assessing Swallowing Function After Transoral Robotic Surgery (TORS) for Head and Neck Cancer
Brief Title: Modified Barium Swallow in Measuring Swallowing Function After Surgery in Patients With Oropharyngeal Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to secure funding.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCCWFU 97312; NCI-2012-02165 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA012197 (NIH)
Record Dates: First submitted 2013-01-11; First posted 2013-01-15 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Oropharyngeal Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (modified barium swallow) (Experimental): Patients undergo the modified barium swallow, comprising swallowing boluses of thin liquid barium, barium honey, barium pudding, and barium crackers while undergoing fluoroscopic imaging.
  Interventions: Procedure: diagnostic imaging; Other: questionnaire administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Procedure: diagnostic imaging — Undergo MBS
Other: questionnaire administration — Correlative studies
Procedure: quality-of-life assessment — Correlative studies
  Other Names: quality of life assessment

SUMMARY:
This pilot clinical trial studies the modified barium swallow in measuring swallowing function after surgery in patients with oropharyngeal cancer who have undergone surgery. New diagnostic procedures, such as the modified barium swallow, may be effective in studying the side effects of cancer therapy in patients who received treatment for oropharyngeal cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare aspiration in oropharyngeal carcinoma patients that underwent transoral robotic surgery (TORS) vs. chemoradiotherapy (CRT) via an objective instrument, the modified barium swallow (MBS).

SECONDARY OBJECTIVES:

I. To compare patient-perceived swallowing function of oropharyngeal carcinoma patients that underwent TORS vs. CRT via a subjective instrument, the M.D. Anderson Dysphagia Inventory (MDADI) using the total MDADI score.

II. To compare patient-perceived swallowing function of oropharyngeal carcinoma patients that underwent TORS vs. CRT via a second subjective instrument, the Eating Assessment Tool (EAT-10) using the total EAT-10 score.

III. To estimate the correlation between the maximum Penetration Aspiration Scale (PAS) score and MDADI total score in TORS or CRT oropharyngeal carcinoma patients regardless of treatment modality.

IV. To estimate the correlation between the maximum PAS score and EAT-10 total score in TORS or CRT oropharyngeal carcinoma patients regardless of treatment modality.

V. To estimate the correlation between MDADI total score and EAT-10 total score in TORS or CRT oropharyngeal carcinoma patients regardless of treatment modality.

VI. To estimate cervical esophageal stricture diameters after TORS vs. CRT via an objective instrument, the MBS.

OUTLINE:

Patients undergo the modified barium swallow, comprising swallowing boluses of thin liquid barium, barium honey, barium pudding, and barium crackers while undergoing fluoroscopic imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have undergone TORS or CRT for oropharyngeal carcinoma 6-24 months prior at Wake Forest University Baptist Hospital (WFUBH)
* In CRT treated participants, CRT had to be delivered as a primary modality with curative intent
* In TORS treated participants, TORS had to be done as a primary modality with curative intent
* Written informed consent
* No evidence of recurrent disease or second primary tumors on physical examination

Exclusion Criteria:

* Previous head and neck surgery, radiation, or chemotherapy preceding TORS
* Previous head and neck surgery preceding CRT
* If CRT patient, candidacy for TORS is not met
* Known neurologic dysfunction affecting swallowing
* Evidence of recurrent or second primary cancers on examination
* Patient pregnancy (due to radiation exposure risk to unborn fetus)
* Inability to grant informed consent

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Dichotomized aspiration, measured via the maximum Penetration-Aspiration Scale (PAS) delineated from the MBS | Baseline
  The maximum PAS score will be dichotomized into aspiration vs no aspiration. The highest (closest to 8 on the PAS scale) PAS score of the 10 swallows will be used for dichotomization. A PAS score of 6 or greater indicates aspiration, while a PAS score of 5 or less is indicative of no aspiration. McNemar's test for correlated proportions will be used to assess the difference between the two treatment groups.

SECONDARY OUTCOMES:
Swallowing function, assessed by the MDADI score | Baseline
  The total MDADI score will be analyzed using paired t-tests.
Perceived subjective swallowing function, assessed using the EAT-10 | Baseline
  The total EAT-10 score will be analyzed using paired t-tests.
Cervical esophageal stricture measurements | Baseline
  A paired t-test will be used to assess the difference in cervical esophageal stricture diameters between the two treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Waltonen, Principal Investigator — Wake Forest University Health Sciences